CLINICAL TRIAL: NCT05423236
Title: Clinical Characteristics of Lung Cancer in China: 8-Year Population-Based Study
Brief Title: Clinical Characteristics of Lung Cancer in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Yayi He, Principal Investigator, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 2022LY0414
Record Dates: First submitted 2022-05-12; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Lung Cancer
Keywords: Cross-sectional Study; Clinical Characteristics
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a single-center, real-world and large-population-based retrospective study. In the current study, the investigators not only describe the changes of demographic and basic clinicopathological characteristics of lung cancer during recent years but delineate the correlation between clinicopathological features and common clinical blood tests in such a large population.

DETAILED DESCRIPTION:
In this study, the investigators will collected all lung cancer patients diagnosed in Shanghai Pulmonary Hospital from 2012 to 2020. By conducting this population based study, the investigators would like to delineate changes of characteristics of lung cancer in Chinese patients during these years. Meanwhile, the investigators will compare clinicopathological features, routine blood tests, blood biochemical tests and coagulation status among participants at different stages. This comparing will assist the investigators to understand systemic changes during lung cancer progression. The same comparison will also be conducted among participants having different driver mutation through which the investigators will further understand the characteristics of different patients and treat patients more precisely.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have medical records in our hospital.
2. Patients were diagnosed as lung cancer by pathological examination.

Exclusion Criteria:

1. Patients were lack of accurate pathological diagnoses.
2. Pathological diagnosis was benign disease or metastatic cancer from other organs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population was patient who was diagnosed as lung cancer at Shanghai Pulmonary Hospital from January 1st, 2012 to October 31st, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 119785 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Comprehensive analysis of clinical characteristics of lung cancer of all participants | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The changes of demographic characteristics and clinicopathological characteristics of Chinese lung cancer patients during the 8 years, from 2012 to 2020, will be analyzed.
Measurement of prothrombin time (PT) would be performed in all participants | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The investigators collected the prothrombin time (PT) (the unit is second). Then the investigators would compare PT among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.
Measurement of activated partial thromboplastin time (APTT) would be performed in all participants | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The investigators collected the activated partial thromboplastin time (APTT) (the unit is second). Then the investigators would compare APTT among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.
Measurement of thrombin time (TT) would be performed in all participants | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The investigators collected the thrombin time (TT) (the unit is second). Then the investigators would compare TT among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.
Measurement of fibrinogen would be performed in all participants | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The investigators collected the blood fibrinogen content (the unit is gram per liter). Then the investigators would compare blood fibrinogen content among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.
Measurement of D-dimer would be performed in all participants | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The investigators collected the blood D-dimer content (the unit is nanogram per milliliter). Then the investigators would compare blood D-dimer content among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.
Measurement of fibrinogen degradation product (FDP) would be performed in all participants | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The investigators collected the blood fibrinogen degradation product (FDP) (the unit is microgram per milliliter). Then the investigators would compare blood FDP content among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.
Complete blood cell count (CBC) would be performed in all participants | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The investigators collected the result of complete blood cell count (CBC) of all participants. Then the investigators would compare CBC results among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.
Renal function test would be performed in all participants | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The investigators collected the result of creatinine (the unit is micromole per liter) of all participants. Then the investigators would compare creatinine level among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.
Alanine aminotransferase would be measured in all participants | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The results of measurement of alanine aminotransferase (ALT) (the unit is unit per liter) would be collected. Then the investigators would compare ALT among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.
Aspartate aminotransferase would be measured in all participants | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The results of measurement of aspartate aminotransferase (AST) (the unit is unit per liter) would be collected. Then the investigators would compare AST among the participants having different driver mutation. Meanwhile, these would also be compared among the participants at different stage.
Alkaline phosphatase would be measured in all participants | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The results of measurement of alkaline phosphatase (ALP) (the unit is unit per liter) would be collected. Then the investigators would compare ALP among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.
Gamma-glutamyl transferase would be measured in all participants | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The results of measurement of gamma-glutamyl transferase (GGT) (the unit is unit per liter) would be collected. Then the investigators would compare GGT among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.

SECONDARY OUTCOMES:
Blood electrolyte level would be tested | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The investigators collected the result of sodium, potassium, calcium, chloride, phosphate and magnesium (the unit is millimole per liter) of all participants. Then the investigators would compare these among the participants having different driver mutation. Meanwhile, these would also be compared among the participants at different stage.
Measurement of total glycerol would be performed | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The investigators collected the result of total glycerol (the unit is millimole per liter) of participants. Then the investigators would compare it among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.
Measurement of total cholesterol would be performed | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The investigators collected the result of total cholesterol (the unit is micromole per liter) of participants. Then the investigators would compare it among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.
Measurement of low density lipoprotein cholesterol (LDL-C) would be performed | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The investigators collected the result of LDL-C (the unit is millimole per liter) of participants. Then the investigators would compare it among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.
Measurement of high density lipoprotein cholesterol (HDL-C) would be performed | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The investigators collected the result of HDL-C (the unit is millimole per liter) of participants. Then the investigators would compare it among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.
Fasting blood glucose (FBG) test would be performed | The data will be collected from medical records in recent 8 years from 2012 to 2020. And investigators will analyze these data in the following 1 year.
  The investigators collected the result of FBG (the unit is millimole per liter) of participants. Then the investigators would compare it among the participants having different driver mutation. Meanwhile, it would also be compared among the participants at different stage.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Result] Al-Samkari H, Leiva O, Dagogo-Jack I, Shaw A, Lennerz J, Iafrate AJ, Bendapudi PK, Connors JM. Impact of ALK Rearrangement on Venous and Arterial Thrombotic Risk in NSCLC. J Thorac Oncol. 2020 Sep;15(9):1497-1506. doi: 10.1016/j.jtho.2020.04.033. Epub 2020 May 11. PMID 32437899
- [Result] Roopkumar J, Poudel SK, Gervaso L, Reddy CA, Velcheti V, Pennell NA, McCrae KR, Khorana AA. Risk of thromboembolism in patients with ALK- and EGFR-mutant lung cancer: A cohort study. J Thromb Haemost. 2021 Mar;19(3):822-829. doi: 10.1111/jth.15215. Epub 2021 Jan 24. PMID 33314597
- [Result] Zhu VW, Zhao JJ, Gao Y, Syn NL, Zhang SS, Ou SI, Bauer KA, Nagasaka M. Thromboembolism in ALK+ and ROS1+ NSCLC patients: A systematic review and meta-analysis. Lung Cancer. 2021 Jul;157:147-155. doi: 10.1016/j.lungcan.2021.05.019. Epub 2021 May 20. PMID 34049720
- [Result] Qian X, Fu M, Zheng J, Zhou J, Zhou J. Driver Genes Associated With the Incidence of Venous Thromboembolism in Patients With Non-Small-Cell Lung Cancer: A Systematic Review and Meta-Analysis. Front Oncol. 2021 Apr 29;11:680191. doi: 10.3389/fonc.2021.680191. eCollection 2021. PMID 33996610
- [Derived] Xu K, Wang H, Li S, Zhao L, Liu X, Liu Y, Ye L, Liu X, Li L, He Y. Changing profile of lung cancer clinical characteristics in China: Over 8-year population-based study. Chin Med J Pulm Crit Care Med. 2023 Sep 15;1(3):188-194. doi: 10.1016/j.pccm.2023.08.006. eCollection 2023 Sep. PMID 39171125